CLINICAL TRIAL: NCT06128837
Title: A Multicenter, Randomized, Open-label, Parallel-design Phase 3 Study to Evaluate the Efficacy and Safety of LY01610 (Irinotecan Hydrochloride Liposome Injection) Versus Topotecan in Patients With Recurrent Small Cell Lung Cancer (SCLC)
Brief Title: Study of LY01610 in Patients With Recurrent Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY01610/CT-CHN-304
Record Dates: First submitted 2023-10-18; First posted 2023-11-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Relapsed Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01610 (Experimental): Patients will consecutively receive LY01610 on Day 1 q2wk (every two weeks = one treatment cycle)
  Interventions: Drug: Irinotecan hydrochloride liposome Injection
- Topotecan (Active Comparator): Patients will consecutively receive Topotecan on Days 1-5 q3wk(every three weeks = one treatment cycle)
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Irinotecan hydrochloride liposome Injection — Irinotecan hydrochloride liposome Injection 80 mg/m² intravenously Days 1 q2wk
  Arms: LY01610
Drug: Topotecan — Topotecan 1.2 mg/m² intravenously Days 1-5 q3w
  Arms: Topotecan

SUMMARY:
This is a multicenter，randomized, open label, active-controlled, parallel-group study comparing efficacy and safety of LY01610(Irinotecan hydrochloride liposome Injection) and Topotecan in Patients with Recurrent Small Cell Lung Cancer (SCLC)

DETAILED DESCRIPTION:
A multicenter, randomized, open-label, parallel study was designed to evaluate the efficacy and safety of LY01610 versus topotecan in the second-line treatment of patients with recurrent SCLC who were diagnosed by histopathology and/or cytology and had disease progression after first-line platinum-based chemotherapy, to conduct a population pharmacokinetics (PopPk) study, and to explore the effect of genetic polymorphisms on the pharmacokinetics properties, efficacy and safety of this product.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female;
2. Patients with histologically and/or cytologically confirmed small cell lung cancer;
3. Disease progression (CTFI ≥ 30 days and ≤ 6 months) occurred after at least 4 cycles of first-line etoposide + platinum two-drug chemotherapy-based treatment, regardless of whether the primary tumor was treated with radiotherapy; the stage of patients with limited stage SCLC should meet more than T1-2, N0, or not suitable for surgery;
4. At least one evaluable lesion (according to RECIST 1.1 criteria);
5. Expected survival time ≥ 3 months;
6. Eastern Cooperative Oncology Group (ECOG) score < 2;
7. Patients who received no liver metastasis; or the number of liver metastases was ≤ 3 and the longest diameter of a single lesion was ≤ 1.5 cm; or although the longest diameter of a single lesion was > 1.5 cm, the imaging was stable for at least 3 weeks after local treatment control;
8. Patients with brain metastasis at baseline should meet all the following conditions: lesions not involving the brainstem, the number of brain metastases ≤ 2 (but patients with only intracranial target lesions should be excluded), imaging stability for at least 3 weeks after local treatment control, and no application of dehydration drugs and hormones before screening,Without any symptoms of brain metastasis;
9. Organ function meeting the following criteria at screening: a.Blood routine: neutrophil (ANC) ≥ 1.5 × 109/L, platelet (PLT) ≥ 100 × 109/L, hemoglobin (Hb) ≥ 90 g/L; b.Liver function: total bilirubin (TBIL) ≤ 1.0 × upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.0 × ULN; if liver metastases, AST and ALT ≤ 3 × ULN; serum albumin ≥ 30 g/L; c.Renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 40 mL/min; d.Coagulation function: Prothrombin time - international normalized ratio (PT-INR) < 1.5;
10. Has fully understood and voluntarily signed a written informed consent form for this study and is able to comply with the requirements and restrictions listed in the informed consent form;
11. Female subjects of childbearing potential and male subjects with partners of childbearing potential agree to use reliable contraceptive measures during the study and within 6 months after the infusion of study drug.

Exclusion Criteria:

1. Pathological diagnosis of compound small cell lung cancer;
2. Patients with meningeal metastasis, spinal cord tumor invasion, spinal cord compression syndrome;
3. Superior vena cava syndrome with symptoms or significantly aggravated imaging, which may require radiotherapy/surgery/endoscopic therapy/intervention and other non-medical treatment; the presence of large amount of pleural effusion, ascites and/or pericardial effusion with local treatment and unstable control;
4. Active infection (including tuberculosis infection) requiring systemic anti-bacterial, antifungal, antiviral and other treatments during screening;
5. Recurrent symptomatic poorly controlled chronic obstructive pulmonary disease, extensive interstitial lung disease (including interstitial pneumonia, pulmonary interstitial fibrosis, etc.) at screening,
6. Extensive radiation pneumonitis, pulmonary embolism or active massive hemoptysis; Patients with severe gastrointestinal diseases or gastrointestinal disorders (such as gastrointestinal bleeding, gastrointestinal obstruction, unhealed peptic ulcer, immune enteritis, ulcerative colitis, Crohn's disease, ischemic necrotizing enteritis, diarrhea > grade 1, other gastrointestinal diseases that may affect the tolerance of chemotherapy) at screening;
7. Patients with the following cardiovascular and cerebrovascular diseases or history:

   1. patients with unstable hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) or a history of hypertensive crisis or hypertensive encephalopathy;
   2. patients with unstable severe arrhythmia;
   3. patients with the following cardiovascular and cerebrovascular diseases within 6 months: myocardial infarction, unstable angina, coronary revascularization/angioplasty, coronary artery bypass grafting, coronary artery stenting, New York Heart Association (NYHA) class ≥ 2 cardiac insufficiency, severe unstable arrhythmia, deep vein thrombosis, pulmonary embolism history, active cerebral infarction, active cerebral hemorrhage;
8. Patients with any of the following conditions:

   1. positive hepatitis B virus surface antigen (HBsAg) test,And peripheral blood hepatitis B virus deoxyribonucleic acid (HBV-DNA) detection ≥ 1000 IU/mL;
   2. hepatitis C virus antibody (HCV-Ab) positive, and hepatitis C virus ribonucleic acid (HCV-RNA) detection ≥ 100 IU/mL;
   3. human immunodeficiency virus antibody (HIV-Ab) detection positive;
9. Other malignancies within 5 years before screening (except cured stage IB or lower cervical cancer, non-invasive basal cell, scale-cell skin cancer or resectable carcinoma in situ);
10. Patients with primary diseases of other important organs (such as nervous system, cardiovascular and cerebrovascular system, urinary system, digestive system, respiratory system or metabolic endocrine system diseases) and the researchers believe that it is not suitable for participants, or for other reasons the researchers believe that it is not suitable for participants;
11. Previous treatment with irinotecan or irinotecan modified, topotecan or other topoisomerase I inhibitors;
12. Known hypersensitivity to irinotecan hydrochloride liposomes or its excipients, structurally similar compounds (such as camptothecin compounds), other liposomal drugs, and topotecan;
13. Those who have been vaccinated with live vaccine or live attenuated vaccine before screening;
14. Patients who have received systemic anti-tumor therapy in 4 weeks before randomization;
15. Patients who have applied other clinical trial drugs/devices before randomization;
16. Patients who have used strong inducers or strong inhibitors of CYP3A4 and strong inhibitors of UGT1A1 before randomization;
17. Adverse reactions caused by previous anti-tumor treatment are not recovered to grade 1 or lower (except alopecia and peripheral neuropathy);
18. History of drug abuse, drug abuse and/or alcoholism;
19. Pregnant or lactating women;
20. Other conditions (including but not limited to unstable nervous system diseases and mental disorders) that are considered unsuitable for inclusion in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death or last contact, whichever occurs first, assessed up to 52 month
  Overall survival is defined as the time from randomization to date of death.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization to the date of progressive disease, death or last tumor assessment or further anticancer treatment, whichever occurs first, assessed up to 52 months
  Progression-free survival is the time from randomization to the first documented objective disease progression (PD) using RECIST v1.1 or death due to any cause, whichever occurs first
Overall response rate | At baseline and every six weeks (± one week) through study completion, an average of 1 year
  Overall response rate (ORR) will be the best response obtained in any evaluation according to RECIST v.1.1
Overall survival rate at 1 year | At 12 months
  Overall survival rate at 1 year is defined as the percentage of people who are still alive at 12 months after randomization.
Duration of response | From the date of first documentation of complete or partial response to the date of documented progression disease, death or last contact, whichever occurs first, assessed up to 52 months
  Duration of response (DoR) will be calculated from the date of first documentation of response per RECIST v.1.1 (complete or partial response, whichever occurs first) to the date of documented PD or death
Patient-reported outcomes | At baseline and every six weeks (± one week) through study completion, an average of 1 year
  To measure the quality of life of patients, EORTC QLQ-C30/LC13 questionnaire will be analyzed
Maximum plasma concentration | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2（each Cycle is 14 days）
  Maximum plasma concentration of total Irinotecan，free Irinotecan ，and its metabolite SN-38，SN-38G (Cmax) in 20~24 subjects treated with LY01610
Time to maximum plasma concentration | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2（each Cycle is 14 days）
  Time to maximum plasma concentration of total Irinotecan，free Irinotecan ，and its metabolite SN-38，SN-38G (Tmax) in 20~24 subjects treated with LY01610
Area under the plasma concentration-time curve | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2（each Cycle is 14 days）
  Area under the plasma concentration-time curve of total Irinotecan，free Irinotecan ，and its metabolite SN-38，SN-38G (AUC) in 20~24 subjects treated with LY01610
Elimination half-life | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2（each Cycle is 14 days）
  Elimination half-life of total Irinotecan，free Irinotecan，and its metabolite SN-38，SN-38G (t1/2) in 20~24 subjects treated with LY01610
Plasma concentrations for Population PK Analyses | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2（each Cycle is 14 days）
  Pharmacokinetic plasma concentration-time data for total Irinotecan，free Irinotecan，and its metabolite SN-38，SN-38G will be analyzed using population pharmacokinetic methods in all subjects treated with LY01610 and identify the effect of covariates on pharmacokinetic parameters in the subject population
Incidence of treatment-emergent adverse events, serious adverse events and laboratory abnormalities | From the date of randomization through study completion, an average of 1 year
  Safety analyses (adverse events and laboratory analyses) will be performed using the safety population, defined as all patients receiving any study drug

CONTACTS AND LOCATIONS:
Overall Officials: yuankai shi, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China